CLINICAL TRIAL: NCT02076451
Title: PHASE 1, OPEN-LABEL STUDY TO ASSESS THE SAFETY AND TOLERABILITY OF DS-8273A IN SUBJECTS WITH ADVANCED SOLID TUMORS OR LYMPHOMAS
Brief Title: Open-label Study of DS-8273a to Assess Its Safety and Tolerability, and Assess Its Pharmacokinetic and Pharmacodynamic Properties in Subjects With Advanced Solid Tumors or Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS8273-A-U101
Record Dates: First submitted 2014-02-25; First posted 2014-03-03 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2016-02

CONDITIONS: Advanced Solid Tumor; Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — DS-8273a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 2 mg/kg DS-8273a (Experimental): 2 mg/kg, 8 mg/kg, 16 mg/kg, and 24 mg/kg of DS-8273a; DS-8273a will be administered as an intravenous (IV) solution. Subjects will receive DS-8273a on Day 1 of a 21 day cycle (once every 3 weeks).
  Interventions: Drug: DS-8273a
- 8 mg/kg DS-8273a (Experimental): 2 mg/kg, 8 mg/kg, 16 mg/kg, and 24 mg/kg of DS-8273a; DS-8273a will be administered as an intravenous (IV) solution. Subjects will receive DS-8273a on Day 1 of a 21 day cycle (once every 3 weeks).
  Interventions: Drug: DS-8273a
- 16 mg/kg of DS-8273a (Experimental): 2 mg/kg, 8 mg/kg, 16 mg/kg, and 24 mg/kg of DS-8273a; DS-8273a will be administered as an intravenous (IV) solution. Subjects will receive DS-8273a on Day 1 of a 21 day cycle (once every 3 weeks).
  Interventions: Drug: DS-8273a
- 24 mg/kg of DS-8273a (Experimental): 2 mg/kg, 8 mg/kg, 16 mg/kg, and 24 mg/kg of DS-8273a; DS-8273a will be administered as an intravenous (IV) solution. Subjects will receive DS-8273a on Day 1 of a 21 day cycle (once every 3 weeks).
  Interventions: Drug: DS-8273a

INTERVENTIONS:
Drug: DS-8273a — DS-8273a will be administered as an intravenous (IV) solution. Subjects will receive DS-8273a on Day 1 of a 21 day cycle (once every 3 weeks

SUMMARY:
This will be a Phase 1, open-label study of DS-8273a to assess its safety and tolerability, identify the Maximum Tolerated Dose and/or Maximum Administered Dose, and assess its properties in subjects with advanced solid tumors or lymphomas.

Up to 5 US sites are planned for participation in Part 1 (Dose Escalation) and Part 2 (Dose Expansion) in subjects with solid tumors or lymphomas.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically or cytologically documented advanced solid tumor or lymphoma that has relapsed from or is refractory to standard treatment, and for whom no standard treatment is available.
* Man or woman >= 18 years old.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Has adequate bone marrow function, defined as: Platelet count >= 100 X 10*9/L Hemoglobin level >= 9.0 g/dL Absolute neutrophil count >= 1.5 x 10*9/L
* Has adequate renal function, defined as: Creatinine clearance >= 60 mL/minute, as calculated using the modified Cockroft Gault equation, ([{140 - age in years} × {actual weight in kg}] divided by [{72 × serum creatinine in mg/dL} multiplied by 0.85 if female]), OR creatinine <= 1.5 X upper limit of normal (ULN)
* Has adequate hepatic function, defined as: AST/ALT <= 3 X ULN (if liver metastases are present, <= 5 X ULN) Bilirubin <= 1.5 X ULN
* Has adequate blood clotting function, defined as: International normalized ratio and activated partial thromboplastin time <= 1.5 X ULN
* Subject should be able to provide written informed consent and comply with protocol visits and procedures.
* Subject (male and female) of childbearing/ reproductive potential must agree to use double barrier contraceptive measures or avoid intercourse during the study and for 90 days after the last dose of study drug.
* Subject must be fully informed about their illness and the investigational nature of the study protocol (including foreseeable risks and possible side effects) and must sign and date an Institutional Review Board-approved Informed Consent Form (including Health Insurance Portability and Accountability Act authorization, if applicable) before performance of any study specific procedures or tests.
* Is willing to provide pre-existing diagnostic or resected tumor samples, such as paraffin-embedded sections. Providing a fresh tumor biopsy sample is optional.
* Following treatment-free period prior to enrollment to the study: i)Surgery: 4 weeks for major surgery (e.g., laparotomy and thoracotomy); 2 weeks for less extensive surgery (e.g., colostomy) ii)Radiation: 4 weeks (2 weeks for palliative irradiation to bone metastases [except for pelvic irradiation], and brain metastasis) iii) Chemotherapy (including systemic treatment with anticancer therapy and retinoid therapy): 3 weeks (6 weeks for nitrosourea antineoplastic agent and mitomycin C) iv) Antibody-based therapy: 4 weeks v) Small molecule targeted agents: If myelosuppression is not expected, 2 weeks or 5 half-lives, whichever is longer; otherwise, 3 weeks vi) Hormonal treatment: 3 weeks. Previous and concurrent use of hormone replacement therapy, the use of gonadotropin-releasing hormone modulators for prostate cancer, and the use of somatostatin analogs for neuroendocrine tumors are permitted if such therapy has not been changed within 8 weeks before study drug treatment. vii) Pleurodesis: 2 weeks

Exclusion Criteria:

* Has a history of primary central nervous system malignancy.
* Has an uncontrolled infection requiring IV antibiotics, antivirals, or antifungals, known human immunodeficiency virus infection, or active hepatitis B or C infection.
* Has received an allogeneic bone marrow or allogeneic stem cell transplant.
* Has a concomitant medical condition that would increase the risk of toxicity, in the opinion of the Investigator or Sponsor.
* Has clinically active brain metastases, defined as untreated and symptomatic, or requiring therapy with steroids or anticonvulsants to control associated symptoms. Subjects with treated brain metastases that are no longer symptomatic and who require no treatment with steroids may be included in the study if they have recovered from the acute toxic effect of radiotherapy. A minimum of 4 weeks must have elapsed between the end of whole brain radiotherapy and study enrollment (2 weeks for stereotactic radiotherapy).
* Has unresolved toxicities from prior anti-cancer therapies, defined as toxicities (chemotherapy, hormonal treatment, radiation, and/or surgery) not yet resolved to NCI-CTCAE, v4, Grade <= 1 or baseline; other than alopecia, skin toxicity (Grade 1), according to NCI-CTCAE, v4. Subjects with chronic Grade 2 toxicities may be eligible per the discretion of the Investigator and Sponsor (e.g., Grade 2 chemotherapy-induced peripheral neuropathy).
* Had an autologous transplant within 3 months of starting study drug treatment.
* Participated in a therapeutic clinical study within 3 weeks (2 weeks or 5 half-lives, whichever is longer, for small-molecule targeted agents) before study drug treatment, or current participation in other therapeutic investigational procedures.
* Prolongation of corrected QT interval by Fridericia's method (QTcF) at rest, where the mean QTcF interval is > 450 ms for males and > 470 ms for females based on triplicate electrocardiogram (ECG).
* Pregnant or breastfeeding.
* Substance abuse or medical, psychological, or social conditions that, in the opinion of the Investigator, may interfere with the subject's participation in the clinical study or evaluation of the clinical study results.
* Prior treatment with a human DR5 agonist.
* Life expectancy < 3 months in the opinion of the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
number of adverse events | 21 days
  To assess the safety and tolerability of DS 8273a in subjects with advanced solid tumors or lymphomas who have relapsed from or are refractory to standard treatment and for whom no standard treatment is available.
maximum tolerated dose | 21 days
  To determine the maximum tolerated dose (MTD) and/or maximum administered dose (MAD), and tentative recommended Phase 2 dose (RP2D) of DS-8273a in subjects with advanced solid tumors or lymphomas.

SECONDARY OUTCOMES:
tumor response | 21 days
  To evaluate the tumor response to DS-8273a using corresponding standard response criteria, Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, or revised International Working Group (IWG) criteria for lymphoma, if applicable.
incidence of human anti-human antibody (HAHA) formation | 21 days
  evaluate the incidence of human anti-human antibody (HAHA) formation
determine the pharmacokinetics of DS-8273a | 21 days
  determine the pharmacokinetics of DS-8273; area under the concentration versus-time curve [AUC], maximum [peak] observed concentration in plasma [Cmax], time of maximum observed concentration [tmax], terminal elimination half-life t1/2.

CONTACTS AND LOCATIONS:
Locations (1):
- Sarah Cannon Research Institute / Tennesee Oncology, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/